CLINICAL TRIAL: NCT00601224
Title: Social Cognition and Interaction Training for Schizophrenia
Brief Title: Social Cognition and Interaction Training for Improving Social Functioning in People With Schizophrenia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Penn, PhD, Professor of Psychology, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R34MH080010 (NIH); R34MH080010 (NIH); DATR A2-AISZ
Record Dates: First submitted 2008-01-15; First posted 2008-01-28 (Estimated); Last update posted 2013-03-29 (Estimated); Status verified 2013-03

CONDITIONS: Schizophrenia
Keywords: Social Cognition; Group Therapy; Psychosocial Intervention
MeSH Terms: conditions — Schizophrenia | interventions — Therapeutics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Participants will receive social cognition and interaction training plus treatment as usual
  Interventions: Behavioral: Social cognition and interaction training (SCIT); Behavioral: Treatment as usual (TAU)
- 2 (Active Comparator): Participants will receive treatment as usual
  Interventions: Behavioral: Treatment as usual (TAU)

INTERVENTIONS:
Behavioral: Social cognition and interaction training (SCIT) — SCIT is a group-based treatment that has the goal of improving social cognition and social functioning for individuals with psychotic disorders. SCIT is composed of three phases: emotion training, figuring out situations, and integration. SCIT will be delivered by two therapists in 20 weekly sessions over 5 months.
  Arms: 1
Behavioral: Treatment as usual (TAU) — TAU will involve routine care and meeting with case-managers and healthcare providers on an as-needed basis.

SUMMARY:
This study will determine the effectiveness of social cognition and interaction training, a manual-based group therapy program, in helping people with schizophrenia improve their social cognition and social functioning.

DETAILED DESCRIPTION:
Schizophrenia is a serious mental condition that affects approximately 1.1% of adults in the United States. People with schizophrenia experience reality perception impairments, which most commonly manifest as hallucinations, extreme paranoia, social withdrawal, and disordered thinking. Deficits in social functioning are a core feature of schizophrenia. In an effort to improve social functioning, there has been growing interest in identifying factors that underlie psychosocial impairments. One such identified factor has been neurocognition, but treatments that target solely cognitive processes do not always help overall social functioning. Social cognition and interaction training (SCIT), a group-based treatment that aims to improve both processing social information and functioning, may be an effective treatment for enhancing the social skills of people with schizophrenia. This study will compare the effectiveness of SCIT versus treatment as usual (TAU) in helping people with schizophrenia improve their social cognition and social functioning.

Participation in this single-blind study will last 11 months. All potential participants will undergo initial screening, involving the completion of a few brief tasks testing social functioning. Eligible participants will then be randomly assigned to receive SCIT plus TAU or TAU alone. Participants assigned to receive SCIT will attend twenty 1-hour weekly group sessions over 5 months. During these sessions, participants will learn ways to manage emotions, work through problems, and integrate into social situations. Participants assigned to TAU alone will meet with their case managers and healthcare provider on an as-needed basis. All participants will undergo assessments of social cognition, social functioning, and psychotic symptoms prior to treatment, immediately post-treatment, and 6 months after treatment. Each assessment will last 3 hours and will include interviews, questionnaires, and a variety of tasks testing social skills. Researchers will also contact a family member or significant other about the participant's social functioning at the same three assessment times noted above.

ELIGIBILITY:
Inclusion Criteria:

* Meets DSM-IV criteria for schizophrenia or schizoaffective disorder, based on the Structured Interview of DSM-IV patient version (SCID-P)

Exclusion Criteria:

* Meets current criteria for substance dependence, based on the SCID-P
* Meets criteria for metal retardation (e.g., has an IQ of less than 80)
* History of brain injuries
* Difficulties interacting with others, based on ratings on items from the Social Functioning Scale that tap interactional skills

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2007-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Face Emotion Identification Task (FEIT) | Measured at baseline, post-treatment, and 6-month follow-up
Face Emotion Discrimination Task (FEDT) | Measured at baseline, post-treatment, and 6-month follow-up
The Hinting Task | Measured at baseline, post-treatment, and 6-month follow-up
The Awareness of Social Inference Test (TASIT) | Measured at baseline, post-treatment, and 6-month follow-up
Ambiguous Intentions Hostility Questionnaire(AIHQ) | Measured at baseline, post-treatment, and 6-month follow-up

SECONDARY OUTCOMES:
"Beads in the Jar" Task | Measured at baseline, post-treatment, and 6-month follow-up
Quality of Life Scale (QLS) | Measured at baseline, post-treatment, and 6-month follow-up
Positive and Negative Syndrome Scale (PANSS) | Measured at baseline, post-treatment, and 6-month follow-up
Social Skills Performance Assessment (SSPA) | Measured at baseline, post-treatment, and 6-month follow-up
Schizophrenia Cognition Rating Scale (SCoRS) | Measured at baseline, post-treatment, and 6-month follow-up
Overt Social Cognition: A Rating Scale (OSCARS) | Measured at baseline, post-treatment, and 6-month follow-up
Lecomte Self-Esteem Scale | Measured at baseline, post-treatment, and 6-month follow-up
Number of Hospital Admissions | Measured at baseline, post-treatment, and 6-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: David L. Penn, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina Hospitals, Chapel Hill, North Carolina, United States